CLINICAL TRIAL: NCT02400541
Title: Prospective Evaluation of Neuropsychological and Clinical Impact of Cognitive Remediation Program Among Children and Adolescents Treated for Anorexia Nervosa
Brief Title: Efficacity of Cognitive Remediation Treatment Compared to a Controlled Group in Young Patient With Anorexia Nervosa
Acronym: RECOGAMEA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P130905
Record Dates: First submitted 2015-01-27; First posted 2015-03-27 (Estimated); Last update posted 2020-04-29 (Actual); Status verified 2020-04

CONDITIONS: Anorexia Nervosa
Keywords: Anorexia nervosa; Cognitive remediation therapy
MeSH Terms: conditions — Anorexia Nervosa | interventions — Relaxation Therapy

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cognitive remediation therapy (Experimental): 10 sessions of the cognitive remediation therapy program conducted during five weeks
  Interventions: Behavioral: Cognitive remediation therapy
- relaxation therapy (Placebo Comparator): 10 relaxation sessions during 5 weeks
  Interventions: Other: relaxation therapy

INTERVENTIONS:
Behavioral: Cognitive remediation therapy — Our scheme comprises 10 biweekly sessions ( 5 in group and 5 single) . Each session last about 45 minutes.
  Individual sessions will be held with the patient and a therapist trained in the CRT; group sessions will be led by two therapists trained in CRT and regroup the maximum 5 patients.
  Arms: Cognitive remediation therapy
Other: relaxation therapy — Our scheme comprises 10 biweekly sessions. Each session last about 45 minutes.
  Arms: relaxation therapy

SUMMARY:
The aim of research is to test in a randomized clinical trial with active sessions, the efficacy of cognitive remediation therapy in children anorexia nervosa compared to a controlled group. The investigators want to confirm the efficacy of cognitive remediation treatment in children's flexibility problems.

DETAILED DESCRIPTION:
In this research, the investigators want to evaluate remediation cognitive therapy in anorexia nervosa compared to a controlled group (relaxation) based on different factors that testified the cognitive improvement of patients: one week after therapy, six months after and one year after.

Those factors are:

Weight, perfectionism and food symptomatology, temperament, therapeutic alliance and change motivation, clinical evolution of anorexia nervosa, self esteem, executive functions, neuropsychological performance (flexibility and central coherence).

ELIGIBILITY:
Inclusion Criteria:

* Pathology

  * DSM IV criteria of restrictive anorexia nervosa (AN- R), but not requiring amenorrhea or DSM V
  * Accepting and their parents to participate in the study ( signed consents )
* Topics

  * Female supported for AN- R
  * Aged 8 to 16 years
  * Fluent French
  * Inpatients or outpatients suffering of restrictive anorexia nervosa
* Treatments

  * Supports standard load ( family psychotherapy , dietary management , medical monitoring )
  * In case of anxiety or depression , patients may receive additional psychotropic prescription which should be mentioned in the record
  * Treatments previously followed by patients and treatments for other conditions should be described

Exclusion Criteria:

* Pathology

  * Mental Retardation
  * Schizophrenia
  * Organic brain disorder ( encephalitis , degenerative brain tumor , cerebral neuro- degenerative disease , multiple sclerosis , amyotrophic lateral sclerosis, epilepsy )
  * Metabolic Pathology interfere with feeding or its regulation
  * Trouble consumption current substance
  * Severe somatic pathology , progressive or likely to be life -threatening
* Topics The subjects are not mastering the French language will not be considered

  * Subjects or parents do not have sufficient capacity for understanding instructions and consent
  * No affiliation in social security ( beneficiary or legal )

Ages: 8 Years to 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Enrollment: 65 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2019-12-22 (Actual); Study Completion 2019-12-22 (Actual)

PRIMARY OUTCOMES:
cognitive flexibility | 6 months after therapy
  behavioral characteristics related to cognitive difficulties flexibility of anorexic patients, as measured in the medium term (6 months post treatment) by the score of the subscale "shift" BRIEF parent version of the scale (BRIEF-PR).

SECONDARY OUTCOMES:
Weight status | 6 months and one year
  Assess the impact of cognitive remediation therapy on :Weight status by the Body Mass Index
Food symptoms and perfectionism | 6 months and one year
  Assess the impact of cognitive remediation therapy on :Food symptoms and perfectionism measured by the Eating Disorders Inventory auto questionnaire, EDI-2
Temperamental profile | 6 months after therapy
  Assess the impact of cognitive remediation therapy on :Temperamental profile measured by the Junior Temperament and Character Inventory questionnaire
Therapeutic alliance and motivation to change | 6 months and one year
  Assess the impact of cognitive remediation therapy on : therapeutic alliance and motivation to change measured by self-reported scales Helping Alliance Questionnaire-11 and MOTIV
Self-esteem | 6 months and one year
  measured by the Rosenberg Self-Esteem Scale
Executive functions | 6 months and one year
  measured by the scale BRIEF-Parent Report
Neuropsychological performance in particular flexibility and central coherence | 6 months and one year
  measured by tests of WCST (Wisconsin Card Sorting Test), Geft (Group Embedded Figure Test) and tests the battery Ravello Profile (Tower, Verbal Fluency Test VFT, Trail Making Test TMT, Rey Complex Figure Test Osterreich ROCFT )

CONTACTS AND LOCATIONS:
Overall Officials: Asch Muriel, PHD, Principal Investigator — -Hôpital Robert Debré, Service de psychiatrie de l'enfant et de l'adolescent
Locations (1):
- Asch, Paris, France